CLINICAL TRIAL: NCT06018727
Title: Role Of Sensitivity to neuroEndocrine Systems in Social Decisions
Acronym: ROSES
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Changed study design and it is no longer a clinical trial.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-1839
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-08

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Hydrocortisone; Yohimbine; Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydrocortisone + Yohimbine (Experimental): Participants will ingest hydrocortisone and yohimbine during Session 2 approximately 10 minutes into the session.
  Interventions: Drug: Hydrocortisone; Dietary Supplement: Yohimbine
- Placebo + Placebo (Placebo Comparator): Participants will orally ingest two placebos during Session 2 approximately 10 minutes into the session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone 20 mg capsule will be administered orally.
  Other Names: Cortef
  Arms: Hydrocortisone + Yohimbine
Dietary Supplement: Yohimbine — Yohimbine 20 mg capsule will be administered orally.
  Other Names: Yohimbine Hydrochloride
  Arms: Hydrocortisone + Yohimbine
Drug: Placebo — Two placebos will be administered orally.
  Other Names: Sugar pill
  Arms: Placebo + Placebo

SUMMARY:
The purpose of this research study is to investigate how personality traits and neuroendocrine systems relate to decision-making patterns in individuals 18-45 years old. The main question it aims to answer is how neuroendocrine activity impacts decision-making.

This study has two components. First, there will be an online session that participants complete to consent into the study, complete self-report surveys and a cognitive assessment, and confirm their eligibility for the second part of the study. If eligible to continue, participants will complete one in-person experiment session, during which they will complete self-report measures and a decision-making task. During the in-person session, participants will be randomly assigned (like flipping a coin) to ingest either a placebo (non-active) or the combination of hydrocortisone and yohimbine.

DETAILED DESCRIPTION:
This study has two components. First, there will be a 60 minute online session. During this session, participants will first be asked to complete the informed consent process, a demographics and contact form, a series of questionnaires, a working memory assessment, and a HIPAA authorization. Researchers will also conduct a brief interview about the participant's medical history (including questions about mood, personality, and symptoms of borderline personality disorder), which is used to assess eligibility for participation in the study.

If eligible to continue, participants will complete one 90 minute in-person experiment session. During the in-person session, participants will be randomly assigned (like flipping a coin) to ingest either a placebo (non-active) or the combination of hydrocortisone and yohimbine. Ingesting hydrocortisone and yohimbine will increase participants' neuroendocrine (hormone) levels, which naturally become elevated in response to stress. After ingesting either the placebo or hydrocortisone plus yohimbine, participants will complete a series of questionnaires on a computer as well as an online decision-making task. While completing the computer task, participants' heart rate and pupil size activity will be monitored using an ECG monitor and an eye tracker. Three salivary samples will also be collected during this session: one immediately before participants ingest the placebo or hydrocortisone/yohimbine combination and two immediately before and after participants complete the computer game. These salivary samples will be collected, stored, then assayed, a process that allows us to measure participants' cortisol levels, a hormone important for the body's stress response.

ELIGIBILITY:
Inclusion Criteria:

Borderline Personality Disorder (BPD) group:

* Score of 38 or higher on PAI-BOR
* Participants in the BPD group will be primarily recruited from the two DEPENd lab studies that maintain large samples of BPD participants. To ensure maximal similarity between BPD participants recruited from other DEPENd lab studies and BPD participants recruited through other recruitment sources, the investigators will use the same criteria for the BPD group in the ROSES study as the criteria used in the other DEPENd lab studies. BPD participants in the two DEPENd lab studies from which the investigators will be recruiting must meet the following criteria:

  1. 3+ BPD symptoms, one of which must be affective instability, per clinical interview
  2. Participants must score at least 80 on the Reynolds Intellectual Screening Test (RIST).

Matched Control (MC) group:

* Score of 12 or lower on PAI-BOR
* Score below 50th percentile on WHODAS

Combined Inclusion Criteria:

* Ages 18-45
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Willingness to participate in all components of the study
* Access to necessary resources for participating in the virtual Session 1 (i.e., computer, smartphone, internet access)
* Participants must be able to speak, understand and read English.
* Participants must have at least 20/40 visual acuity (correct or uncorrected).

Exclusion Criteria:

* Current use of medications that interact adversely with yohimbine

  a. Iobenguane radiopharmaceutical products
* Current use of medications that interact adversely with hydrocortisone

  1. Aldesleukin
  2. Bacillus Calmette-Guérin (BCG) Products
  3. Cladribine
  4. Dengue Tetravalent Vaccine
  5. Desmopressin
  6. Indium 111 Capromab Pendetide
  7. Macimorelin
  8. Mifamurtide
  9. MiFEPRIStone
  10. Natalizumab
  11. Pimecrolimus:
  12. Ruxolitinib (Topical)
  13. Tacrolimus (Topical)
  14. Talimogene Laherparepvec
  15. Tertomotide
  16. Phenytoin
  17. Rifampin
  18. Troleandomycin
  19. Ketoconazole
  20. High-dose aspirin (>30 mg/kg/day)
* Contraindicated medical conditions of yohimbine

  1. Renal dysfunction
  2. Hepatic dysfunction
  3. Heart failure
  4. Psychotic Disorder or psychosis
  5. Hypotension
  6. Diabetes
  7. Heart disease
  8. Kidney disease
  9. Liver disease
  10. Nervous disorder
  11. Gastric ulcer
  12. Duodenal ulcer
* Contraindicated medical conditions of hydrocortisone

  1. Hypersensitivity to hydrocortisone or any component of the formulation
  2. Systemic fungal infections
  3. Latent Tuberculosis, Tuberculosis reactivity, active Tuberculosis
  4. Cardiovascular disease
  5. Diabetes
  6. Gastrointestinal diseases

  i. Diverticulitis ii. Fresh intestinal anastomoses iii. Active or latent peptic ulcer iv. Ulcerative colitis v. Abscess vi. Renal insufficiency vii. Other pyogenic infection g. Hepatic impairment h. Kidney impairment i. Myasthenia gravis j. Osteoporosis k. Pheochromocytoma l. Seizure disorders m. Septic shock or sepsis syndrome n. Systemic sclerosis o. Thyroid disease p. Strongyloides (threadworm) infestation q. Ocular herpes simplex r. Hypertension
* Given a live vaccine within 2 weeks of completing Visit 1. Recent administration of the following vaccines are specifically contraindicated for hydrocortisone:

  1. Typhoid Vaccine
  2. Yellow Fever Vaccine
  3. Poliovirus Vaccine (Live/Trivalent/Oral)
  4. Rubella- or Varicella-Containing Live Vaccines
* Have a current infection
* Pregnancy
* Individuals lactating
* Recent antihypertensive agents
* History of psychotic disorder, Bipolar I disorder, autism spectrum disorder, reactive attachment disorder, pervasive developmental disorder, motor disorder, head injury, mental retardation, neurological disorder, or current substance dependence
* Family history of Bipolar I disorder in a first degree relative.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Goal-directed decision-making in the Social Decision Tree Task (SDTT) | Collected for 30 minutes ~1 hour into Session 2, which takes place on approximately Day 7 of the study
  Measured by choice behavior in SDTT, which is based on the decision tree framework. After each action, participants receive feedback about the effect of that action and the extent to which it added to or took away from their points. If participants make a given choice, the subsequent actions that they can choose are different than if they were to initially make a different choice.
  An action in SDTT is goal-directed if the possible net gain an individual can earn before the end of the current epoch (a "day" in the SDTT) is equal to or higher than the amount they could gain by choosing the alternative action. The investigators will subset trials so that 1 is coded as choosing the immediately valuable action at the expense of the optimal and 0 is coded as choosing the optimal at the expense of the immediately valuable action. This outcome variable is binary. An action is defined as social if it is paired with a visual cue with a face on it and non-social if not.
Change in salivary cortisol | Collected immediately before the drug/placebo administration (~5 minutes into the session) and 45 minutes after the drug/placebo administration (~50 minutes into the session) in Session 2, which takes place on approximately Day 7
  The investigators will collect a saliva sample immediately before participants ingest the drugs (or placebos, if in the control condition). They will collect a second saliva sample 45 minutes after the drug (or placebo) ingestion. They will measure cortisol levels in both samples through an assay. The investigators will calculate the change in salivary cortisol by subtracting the measured cortisol in the first saliva sample (collected pre-drug/placebo ingestion) from the measured cortisol in the second saliva sample (collected 45 minutes after the drug/placebo ingestion). Salivary cortisol is measured as nmol/L. Salivary cortisol expected to generally be below 200 nmol/L.
Pupil diameter during SDTT | Collected for 30 minutes ~1 hour into Session 2, which takes place on approximately Day 7 of the study
  The outcome will be measured using eye tracking technology.

SECONDARY OUTCOMES:
Change in valence, measured via the affect grid | Collected immediately before the first saliva collection in Session 2 (~5 minutes into the session) and 45 minutes after the second saliva collection in Session 2 (~50 minutes into the session), which takes place on approximately Day 7
  Change in valence will be assessed through the affect grid. Participants will be presented with a 9x9 grid. The vertical dimension of the grid represents arousal, while horizontal dimension of the grid represents valence. The left side of the grid represents negative valence and the right side represents positive valence. Participants will click a square on the grid with their computer mouse to indicate their current affect. Their valence will be measured before the drug/placebo ingestion and 45 minutes after the drug/placebo administration. The minimum valence score is -4, representing extreme negative valence, and the maximum valence score is 4, representing extreme positive valence. The largest change in valence value is 8 (the maximum positive change in valence from time point 1 to time point 2). The smallest change in valence value is -8 (the maximum negative change in valence from time point 1 to time point 2). If no change in valence, the score will be 0.
Change in arousal, measured via the affect grid | Collected immediately before the first saliva collection in Session 2 (~5 minutes into the session) and 45 minutes after the second saliva collection in Session 2 (~50 minutes into the session), which takes place on approximately Day 7
  Change in arousal will be assessed through the affect grid. Participants will be presented with a 9x9 grid. The vertical dimension of the grid represents arousal, while horizontal dimension of the grid represents valence. The top of the grid represents high arousal and the bottom represents low arousal. Participants will click a square on the grid with their computer mouse to indicate their current affect. Their arousal will be measured before the drug/placebo ingestion and 45 minutes after the drug/placebo administration. The minimum arousal score is -4, representing extremely low arousal, and the maximum arousal score is 4, representing extremely high arousal. The largest change in arousal value is 8 (the maximum positive change in arousal from time point 1 to time point 2). The smallest change in arousal value is -8 (the maximum negative change in arousal from time point 1 to time point 2). If no change in arousal, the score would be 0.
Change in stress, measured via the subjective stress scale | Collected immediately before the first saliva collection in Session 2 (~5 minutes into the session) and 45 minutes after the second saliva collection in Session 2 (~50 minutes into the session), which takes place on approximately Day 7
  Will be assessed via self-report using the one-item subjective stress scale. The scale ranges from 0 to 10. High values indicate more stress, whereas low values indicate less stress.

OTHER OUTCOMES:
Personality Assessment Inventory-Borderline Scale (PAI-BOR) score | Session 1, which takes place on Day 0
  The PAI-BOR measures the number of borderline personality disorder (BPD) symptoms an individual has. The maximum PAI-BOR score is 72, while the minimum score is 0. Lower scores indicate fewer BPD symptoms, whereas higher scores indicate more BPD symptoms.
  The PAI-BOR has five subscales measuring four core BPD traits: Affective Instability, Identity Problems, Negative Relationships, and Self-Harm. The scoring of the subscales are as followed (R = item is reverse-scored): Affective Instability: 1, 4, 7R, 10, 14R, 18; Identity Problems: 2, 5, 8, 11, 15, 19R; Negative Relationships: 3, 6, 9, 12R, 16, 20R; Self-Harm: 13, 17, 21, 22, 23, 24R. The minimum score is 0 and the maximum score is 18 for each of these subscales.
  Individuals in the BPD group must have a PAI-BOR score of 38 or higher. Individuals in the matched control (MC) group must score 12 or lower on the PAI-BOR.
Interbeat Interval (IBI) time series during SDTT | Collected approximately 1 hour into Session 2 for 30 minutes (which takes place on approximately Day 7)
  The time (in milliseconds) between heartbeats. The IBI will be measured using an electrocardiogram (ECG).
Heart rate variability (HRV) during SDTT | Collected approximately 1 hour into Session 2 for 30 minutes (which takes place on approximately Day 7)
  The variation over time of heart beat intervals. HRV will be measured using an electrocardiogram (ECG).
Electrodermal activity (EDA) during SDTT | Collected approximately 1 hour into Session 2 for 30 minutes (which takes place on approximately Day 7)
  Tonic electrodermal activity, which will be determined by using a continuous decomposition analysis.
Skin conductance response during SDTT | Collected approximately 1 hour into Session 2 for 30 minutes (which takes place on approximately Day 7)
  Will be assessed using a skin response module. The skin conductance response will be determined by using a continuous decomposition analysis.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) score | Session 1, which takes place on Day 0
  The WHODAS measures impairment resulting from mental health problems. Participants will complete the 12-item version of the WHODAS. The maximum WHODAS score is 48. The minimum WHODAS score is 0. Lower scores indicate less impairment, whereas higher scores indicate greater impairment.
  Individuals in the matched control (MC) group must have a WHODAS score of 0.
Working memory, assessed by the digit span score | Session 1, which takes place on Day 0
  Working memory will be assessed through the digit span task, where participants are presented with a sequence of numbers containing 3 to 16 numbers. Digit span scores are calculated from the largest number sequence a participant could recall before making two consecutive errors. The minimum score is 3, and the maximum score is 16. Higher scores indicate greater working memory capacity, whereas lower scores indicate lower working memory capacity.
Big Five Inventory (BFI-II) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The Big Five Inventory (BFI-II) measures personality traits via a 60-item questionnaire. These items are measured using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
  There are five domain scales (R = item is reverse-coded): Extraversion, Agreeableness, Conscientiousness, Negative Emotionality, and Openness. The minimum score is 12 while the maximum is 60 for each domain scale.
  The facet scales are Sociability, Assertiveness, Energy Level, Compassion, Respectfulness, Trust, Organization, Productiveness, Responsibility, Anxiety, Depression, Emotional Volatility, Intellectual Curiosity, Aesthetic Sensitivity, and Creative Imagination. The minimum score is 4 while the maximum is 20 for each facet scale.
  Individuals who score high on the BFI-II tend to exhibit more qualities associated with each of the personality traits.
Inventory of Interpersonal Problems (IIP-90) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The Inventory of Interpersonal Problems (IIP-90) is a 90-item questionnaire assessing interpersonal problems. The items are measured using a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). Higher scores indicate more interpersonal problems, whereas lower scores indicate fewer interpersonal problems. The investigators will score each of the eight octant sub scales of the IIP and compute the elevation, dominance, affiliation, and personality disorder subscales on the IIP. Scale scores range from 0 (no interpersonal problems) to 4 (many interpersonal problems).
Traumatic Life Events Questionnaire (TLEQ) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The Traumatic Life Events Questionnaire (TLEQ) measures the amount of exposure an individual has had to potentially traumatic life events. In the first 22 items, participants will be asked how many times they have experienced a certain traumatic event, and will respond with "Never", "Once", "Twice", "3 Times", "4 Times", "5 Times", and "> 5 times". If more than 5 times, they would specify the number of times they experienced the event. The number of times they experienced an event is their score for that item. Item 23 asks which traumatic event that they experienced, if any, causes them the most distress; they will then be asked how much distress that event currently causes them on a 5-point Likert scale ranging from 0 (no distress) to 5 (extreme distress). Total score on TLEQ is the summed score across items assessing experience of different stressful life events. Scores range from 0 (No stressors experienced) to 110 (every stressor experienced 5+ times).
Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior (UPPS-P) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The UPPS-P Impulsive Behavior Scale is a 59-item questionnaire that measures the factors that could lead to impulsive behaviors. Each item is scored on a 4-point Likert scale ranging from 1 (Agree Strongly) to 4 (Disagree Strongly). The minimum score is 59, and the maximum score is 236.
  There are 5 subscales (R = item is reverse-coded): Negative Urgency (2R, 7R, 12R, 17R, 22R, 29R, 34R, 39R, 44R, 50R, 53, 58R), Positive Urgency (5R, 10R, 15R, 20R, 25R, 30R, 35R, 40R, 45R, 49R, 52R, 54R, 57R, 59R), Lack of Premeditation (1, 6, 11, 16, 21, 28, 33, 38, 43, 48, 55), Lack of Perseverance (4, 9R, 14, 19, 24, 27, 32, 37, 42, 47R), and Sensation Seeking (3R, 8R, 13R, 18R, 23R, 26R, 31R, 36R, 41R, 46R, 51R, 56R).
Drug Use Disorders Identification Test (DUDIT) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The Drug Use Disorders Identification Test (DUDIT) is an 11-item questionnaire that measures drug dependence. Higher scores indicate higher drug dependence, whereas lower scores indicate less drug dependence. The first 9 items are scored on a 5-point Likert scale ranging from 0 to 4. The last two questions are scored with 0 (No), 2 (Yes, but not in the past year), or 3 (Yes, during the past year). The minimum score is 0, while the maximum score is 42.
Patient-Reported Outcomes Measurement Information System (PROMIS) Severity of Substance Use (Past 3 months) - Calibrated Items | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The PROMIS Severity of Substance Use (Past 3 months) is a 38-item questionnaire assessing the severity of a participant's substance use. The first question is scored as 1 (No) or 2 (Yes). The following 37 items are a 5-point Likert scale ranging from 1 (Never) to 5 (Almost Always). The researchers will obtain the T-score of the total PROMIS score. Higher scores indicate a higher severity of substance use.
Alcohol Use Disorders Identification Test (AUDIT) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The Alcohol Use Disorders Identification Test (AUDIT) is an 10-item questionnaire that measures alcohol dependence. Higher scores indicate higher alcohol dependence, whereas lower scores indicate less alcohol dependence. The first 8 items are scored on a 5-point Likert scale ranging from 0 to 4. The last two questions are scored with 0 (No), 2 (Yes, but not in the past year), or 4 (Yes, during the past year). The minimum score is 0, while the maximum score is 40.
Personality Inventory for DSM-5 Faceted Brief Form (PID-5-FBF) Score | Collected for 45 minutes after the drug/placebo administration in Session 2 (beginning ~10 minutes into the session), which takes place on approximately Day 7
  The Personality Inventory for DSM-5 (PID-5) is a 100-item questionnaire about characteristics participants may have. The items are measured using a 4-point Likert scale ranging from 0 (Very False/Often False) to 3 (Very True/Often True). The minimum score is 0. The maximum score is 300.
  Facet Scales are Anhedonia, Anxiousness, Attention Seeking, Callousness, Deceitfulness, Depressivity, Distractibility, Eccentricity, Emotional Lability, Grandiosity, Hostility, Impulsivity, Intimacy Avoidance, Irresponsibility, Manipulativeness, Perceptual Dysregulation, Perseveration, Restricted Affectivity, Rigid Perfectionism, Risk Taking, Separation Insecurity, Submissiveness, Suspiciousness, Unusual Beliefs and Experiences, and Withdrawal. Individuals with higher scores exhibit more qualities associated with the facet.
  Domain Scales are Negative Affect, Detachment, Antagonism, Disinhibition, and Psychoticism. Individuals with higher scores exhibit more qualities associated with the domain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Hallquist, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Huys QJ, Eshel N, O'Nions E, Sheridan L, Dayan P, Roiser JP. Bonsai trees in your head: how the pavlovian system sculpts goal-directed choices by pruning decision trees. PLoS Comput Biol. 2012;8(3):e1002410. doi: 10.1371/journal.pcbi.1002410. Epub 2012 Mar 8. PMID 22412360